CLINICAL TRIAL: NCT04334993
Title: A Phase 2, Multicenter, Single Arm Trial to Assess the Safety and Efficacy of a Pediatric Approach to for Young Adults With Acute Lymphoblastic Leukemia With Blinatumomab Therapy for High-risk Patients Prior to Allogeneic Transplantation
Brief Title: Pediatric-type Therapy With Pre-transplant Blinatumomab for HR Patients - Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Israeli Medical Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AYA001
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2020-08

CONDITIONS: Philadelphia-Negative ALL; High-Risk Cancer
Keywords: Philadelphia-Negative ALL; Pediatric therapy; Blinatumomab; Allogeneic transplantation
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Intervention Model Description: This is a national, multicenter, phase II clinical trial
Masking Description: NR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab pre-transplant to high risk Ph-negative ALL pts. (Experimental): Patients designated high risk based on protocol will receive 2 cycles of therapy followed by allogeneic transplantation. Patients ≥45 kg (fixed dose): Cycles 1 and 2: 28 mcg daily administered as a continuous infusion on days 1 to 28 of a 6-week treatment cycle.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Patients with high risk disease features after 2 induction blocks as defined per protocol will be treated with CNS directed block followed by up to 2 cycles of blinatumomab (for B-cell ALL) followed by allogeneic stem cell transplantation.
  Other Names: AIEOP-BFM 2009 protocol - multiagent chemothertapy protocol backbone

SUMMARY:
Despite recent therapeutic advancements, the outcome of young adults with Philadelphia-negative (Ph-neg) acute lymphoblastic leukemia (ALL) and lymphoblastic lymphoma (LBL) remains unsatisfactory, especially in those patients with high-risk disease features. In young adults pediatric-based chemotherapy approaches improve outcome. Furthermore, there is evidence that pre-transplant antibody-based therapy may render patients with positive minimal residual disease (MRD+) to an MRD-negative status (MRD-) and that this may be associated with improved post-transplant outcome.

This is prospective study to evaluate the potential benefit of a modified pediatric-based approach in young adults with Ph-neg ALL. Safety and efficacy of pre-transplant antibody-based consolidation in high-risk patients with Ph-neg ALL will be performed.

DETAILED DESCRIPTION:
This is a national, multicenter, phase II clinical trial to evaluate the potential benefit of a modified pediatric-based approach in young adults with Ph-neg ALL. Safety and efficacy of pre-transplant antibody-based consolidation in high-risk patients with Ph-neg ALL will be assessed.

Young-adult patients eligible with Ph-neg ALL, LBL and mixed phenotype acute leukemia (MPAL) will undergo risk stratification and started on the pediatric Italian Association of Pediatric Hematology Oncology-Berlin-Frankfurt-Münster (AIEOP-BFM) 2009 protocol. Patients defined as having non-high-risk disease features (non-HR) as defined by MRD and/or cytogenetic criteria will complete the non-HR chemotherapy arm per protocol. Patients designated as having HR disease features after 2 induction blocks will be treated with CNS directed block followed by up to 2 cycles of blinatumomab (for B-cell ALL) followed by allogeneic stem cell transplantation. All patients will be centrally assessed for MRD and for Ph-like status.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and <30 years of age at the time of signing the informed consent document.
2. Have a documented diagnosis of Ph-neg ALL, LBL or MPAL according to the WHO 2016 classification (appendix I).
3. Females of childbearing potential (FCBP) may participate, providing they meet the following conditions:

   Agree to use at least two effective contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study, and for 3 months following EOT; and have a negative serum or urine pregnancy test (investigator's discretion; sensitivity at least 25 mIU/mL) at screening; and have a negative serum or urine pregnancy test (investigator's discretion) within 72 hours prior to starting study therapy in the treatment phase (note that the screening serum pregnancy test can be used as the test prior to starting study therapy in treatment phase if it is performed within the 72-hour timeframe).
4. Male subjects with a female partner of childbearing potential must agree to the use of at least two physician-approved contraceptive methods throughout the course of the study and should avoid fathering a child during the course of the study and for 3 months following the last dose of study drug.
5. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
6. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Age <18 or over 30 years at the time of signing the informed consent document.
2. Ph-positive disease.
3. Known Human Immunodeficiency Virus (HIV).
4. Known or suspected hypersensitivity to any of the study drugs.
5. Pregnant or lactating females.
6. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
7. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
8. Participation to an investigational drug trial in the last month before randomization.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 2 years
  Measured from the date of entry on study until treatment failure, relapse from CR, or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  Measured from the date of entry on study until until death from any cause
Early death during induction | 60 days
  Death during the first 60 days from entering study from any cause
MRD status | MRD will be assess by PCR after induction I (day 33), after induction II (week 12), after blinatumomab therapy (prior to HSCT) and at days 30 and 100 post alloHSCT.
  MRD status pre- and post-antibody-based therapy

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Rambam Medical Center, Haifa
  - Shaarei Tzedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No
All data will be coded and uploaded to an electronic CRF (red-cap) to manage abnd analyze data